CLINICAL TRIAL: NCT04152681
Title: Effect and Safety of Apatinib on Radiation-Induced Brain Injury: an Open-label, Single-arm, Phase 2 Study.
Brief Title: Effect and Safety of Apatinib on Radiation-Induced Brain Injury
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yamei Tang, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201910200
Record Dates: First submitted 2019-10-22; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Radiation Injuries
Keywords: Apatinib; Radiation-induced brain injury
MeSH Terms: conditions — Radiation Injuries | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned Interventions (Experimental): Apatinib with a dosage of 250mg once daily for 4 weeks, in the absence of unacceptable toxicity or severe deterioration.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib with a dosage of 250mg once daily for 4 weeks, in the absence of unacceptable toxicity or severe deterioration.

SUMMARY:
Purpose: This early phase 2 clinical trial aims to evaluate the therapeutic effects and safety of apatinib in radiation-induced brain injury.

Further study details as provided by Sun Yet-sen Memorial Hospital, Sun Yat-sen University / Yamei Tang.

Primary outcome measure: The proportion of patients with an objective response defined as ≥ 25% reduction in brain edema volume on MR fluid attenuated inversion recovery (FLAIR) images.

DETAILED DESCRIPTION:
The incidence of nasopharyngeal carcinoma (NPC) is high in China especially in southern China. Radiotherapy is the mainstay of therapy for NPC and greatly improves patient survival. Along with promising therapeutic effects, complications such as radiation dermatitis, temporal lobe necrosis, cognitive impairment, and cranial nerve injury are also associated with radiotherapy. Previously, corticosteroids were considered conventional treatment for radiation-induced brain injury (RI). Unfortunately, only 20% patients with early phase RI seem to benefit from corticosteroid treatment. Moreover, the long-term use of steroids is associated with substantial adverse effects. Recently, bevacizumab, an anti-vascular endothelial growth factor (VEGF) recombinant monoclonal antibody, has been introduced as an efficient treatment for RI. However, the risk of severe adverse effects to bevacizumab, e.g. severe hypertension, proteinuria, nasopharyngeal necrosis and bleeding, limits its usage in certain patients with RI. Apatinib mesylate tablet is an oral small molecule tyrosine kinase inhibitor (TKI), which can specifically bind to vascular endothelial growth factor receptor 2 (VEGFR-2) and strongly inhibit neovascularization. Apatinib is currently used as a third-line treatment for advanced gastric cancer. Previous studies and clinical observation showed that apatinib could significantly improve brain injury after radiation, reduce brain tissue exudation and reduce edema. In this study, investigators will discuss the therapeutic effect of apatinib on RI and evaluate its safety through a prospective phase II clinical trial. It is hopeful to explore a new and effective method for the treatment of RI.

Primary objectives: The primary objective of this phase II, open-label, single-arm designed clinical trial is to evaluate the efficacy and safety of apatinib in patients with RI.

OUTLINE: This is a phase II, open-label, single-arm designed clinical trial. Participants are enrolled and administrated with oral apatinib mesylate tablet for 4 weeks.

Arm 1: Participants receive oral apatinib with a dosage of 250mg once daily for 4 weeks, in the absence of unacceptable toxicity or severe deterioration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥35 years;
* Prior radiotherapy for histologically confirmed head and neck cancer ≥12 months prior to study entry;
* Radiographic evidence to support the diagnosis of radiation-induced brain injury without tumor recurrence;
* Estimated life expectancy must be greater than 12 months;
* Routine laboratory studies：Bilirubin ≤ 1.0 × upper limits of normal (ULN)； Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 1.0 × ULN；Creatinine <1.0 × ULN；White-cell count ≥ 4,000 cells per cubic millimeter；Neutrophils count ≥1500 cells per cubic millimeter；Platelets ≥100,000 cells per cubic millimeter；Hemoglobin ≥110 gram per milliliter；Prothrombin time (PT), activated partial thromboplastin time (APTT), international normalized ratio (INR) within the normal ranges；
* With sufficient cognitive function and language skills for communication and completion of study questionnaires;
* Consent the enrollment of the study.

Exclusion Criteria:

* Evidence of tumor metastasis, recurrence, or invasion;
* Current usage of bevacizumab;
* Current usage of glucocorticoids;
* Evidence of very high intracranial pressure that suggests brain hernia and the need for surgery;
* History of psychiatric disease before radiotherapy;
* History of seizures;
* History of arteriosclerotic cardiovascular diseases (ASCVD), e.g. stroke, myocardial infarction, and unstable angina, within 6 months;
* Present or previous history of cardiac arrhythmia;
* New York Heart Association Grade II or greater congestive heart failure;
* Significant vascular disease, e.g. moderate or severe carotid stenosis, aortic aneurysm, and history of aortic dissection;
* Severe infection;
* History of allergy to relevant drugs;
* Pregnancy, lactation, or fertility program in the following 12 months;
* History or current diagnosis of peripheral nerve disease;
* Abnormal liver and renal function;
* Active tuberculosis;
* A previous history of organ transplantation;
* Infection with the human immunodeficiency virus;
* Participation in other experimental studies;
* Subjects with any other condition which in the investigator's judgment might intervene the outcome of the study.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Overall efficacy rate | 4 weeks
  The proportion of patients with an objective response defined as ≥ 25% reduction in brain edema volume on Magnetic Resonance Imaging (MRI) fluid attenuated inversion recovery (FLAIR) images.

SECONDARY OUTCOMES:
Change of brain necrosis | 4 weeks
  The proportion of patients with an objective response of brain necrosis defined as ≥ 25% reduction in the lesion volume of brain enhancement on post-gadolinium T1-weighted MR images.
Change in neurological function | 4 weeks
  The difference value of the Late Effects of Normal Tissue (LENT)-Subjective, Objective, Management, Analytic (SOMA) questionnaire before and after apatinib regimen. Score range: 0-4. The higher scores means worse outcome.
Change in the quality of life | 4 weeks
  The difference value of World Health Organization Quality of Lif (WHOQOL)-Bref scales before and after apatinib regimen.
  Score range:0-100. Higher scores represent better quality of life.
Change of white matter structural connectivity | 4 weeks
  Structural networks were weighted by measures of white matter microstructure of Neurite orientation dispersion and density imaging (NODDI) (fractional anisotropy, neurite density and orientation dispersion index) before and after apatinib regimen.
Change in cognitive function | 4 weeks
  The difference value of Montreal Cognitive Assessment (MoCA) scales before and after apatinib regimen. Score range:0-30. The higher scores represent better cognitive function.
Change in pain intensity | 4 weeks
  The difference value of Numerical rating scale (NRS) before and after apatinib regimen. Score range: 0-10. The higher scores indicate worse pain.

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, M.D., Ph.D., Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Yamei Tang, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided